CLINICAL TRIAL: NCT01166737
Title: A Randomized Multicenter Study to Compare the Efficacy of Additional Tumor Debulking Surgery vs Chemotherapy Alone in Recurrent Platinum-Sensitive Ovarian Cancer
Brief Title: Study Comparing Tumor Debulking Surgery Versus Chemotherapy Alone in Recurrent Platinum-Sensitive Ovarian Cancer
Acronym: DESKTOPIII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AGO Study Group (Other)
Collaborators: ARCAGY/ GINECO GROUP (Other); Grupo Español de Investigación en Cáncer de Ovario (Other); Cancer Research UK (Other); Shanghai Gynecologic Oncology Group (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: AGO-OVAR OP.4 DESKTOP III
Record Dates: First submitted 2010-07-16; First posted 2010-07-21 (Estimated); Last update posted 2022-01-25 (Actual); Status verified 2021-12

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Peritoneal Cavity Cancer
Keywords: Ovarian Cancer; Cancer of the fallopian tube; Primary peritoneal cancer; Recurrent disease; Platinum-sensitive; Surgery; Chemotherapy; Quality of Life; First recurrence of platinum sensitive:; Fallopian Tube Cancer; or Ovarian Cancer; or Peritoneal Cavity Cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Recurrence | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Arm - Chemotherapy only (No Intervention): Chemotherapy for platinum-sensitive Ovarian Cancer can be selected on investigators choice
- Procedure/Surgery (Experimental): Maximum effort cytoreductive surgery
  Interventions: Procedure: Tumor Debulking Surgery (surgery in recurrent ovarian disease)

INTERVENTIONS:
Procedure: Tumor Debulking Surgery (surgery in recurrent ovarian disease) — Surgery for Patients with platinum-sensitive recurrent ovarian cancer with a positive AGO-score predictive for complete tumor resection
  Arms: Procedure/Surgery

SUMMARY:
It is still not clear whether a positive AGO-score just selects patients with less aggressive biologic tumor behavior who as well would have had a positive outcome by chemotherapy only, or , if it is a score selecting patients who really benefit from surgery. Nevertheless, the AGO-score was confirmed to select patients with a less than 30% risk of ending with residual tumor after surgery for recurrent disease. This could avoid including patients into the present surgical protocol who could not benefit from an operationThe goal of this third DESKTOP study is to evaluate in a prospectively randomized multicentre setting, whether maximum effort of cytoreductive surgery followed by platinum based combination chemotherapy can improve overall survival as compared to platinum based combination chemotherapy alone in AGO-score positive patients.

DETAILED DESCRIPTION:
A predictive score identifying patients who might achieve a complete resection is deemed necessary to select the right patients for a prospective trial on cytoreductive surgery in relapsed ovarian cancer.

Study centres are selected due to their surgical experience in ovarian cancer and/or participation in prior surgical trials in this field. Patients who matched eligibility criteria were allocated randomly 1:1 prospectively to cytoreductive surgery followed by platinum based combination chemotherapy or to platinum based combination chemotherapy alone .

ELIGIBILITY:
Inclusion criteria:

* Patients with first recurrence of platinum sensitive, invasive epithelial ovarian-, fallopian tube- or primary peritoneal cancer of any initial stage.
* Progression-free interval of at least 6 months after end of last platinum-containing therapy, or recurrence within 6 months or later after primary surgery if the patient has not received prior chemotherapy in patients with FIGO I. Non cytostatic maintenance therapy not containing platinum will not be considered for this calculation.
* A positive AGO-score. Obligatory requirements for a positive AGO recurrence score in platinum-sensitive disease:

  1. Performance status ECOG 0
  2. No residual tumor after primary surgery (if unknown, alternatively primary FIGO stage I/II). If report from 1st surgery is not available contact study chairman who will decide whether inclusion is possible or not.
  3. Absence of ascites (cut off < 500 ml: radiological or ultrasound estimation)
* Complete resection of the tumor by median laparotomy seems possible
* Patients who have given their signed and written informed consent and their consent to data transmission and -processing.

Exclusion Criteria:

* Patients with non-epithelial tumors as well as borderline tumors.
* Patients without recurrence who are scheduled for diagnostic/second-look surgery or debulking surgery after completion of chemotherapy
* More than one prior chemotherapy
* Patients with second, third, or later recurrence
* Patients with second malignancies who have been treated by laparotomy, as well as other neoplasms, if the treatment might interfere with the treatment of relapsed ovarian cancer or if major impact on prognosis is expected.
* Patients with so-called platinum-refractory tumor, i.e. progression during chemotherapy or recurrence within 6 months after end of former first platinum-containing therapy
* Only palliative surgery planned
* Radiological signs suggesting metastases not accessible to surgical removal (i.e. complete resection is deemed impossible)
* Any concomitant disease not allowing surgery and/or chemotherapy
* Any medical history indicating excessive peri-operative risk
* Any current medication inducing considerable surgical risk (e.g. bleeding: due to oral anticoagulating agents, bevacizumab)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Actual)
Dates: Start 2010-07 (Actual); Primary Completion 2020-01-17 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Overall survival | Approximately 36 months after last patient randomized and observation of 244 events
  in patients with platinum-sensitive recurrent ovarian cancer with a positive AGO Score

SECONDARY OUTCOMES:
Progression free survival | Progression free survival is defined as interval between date of randomization and 2nd relapse/progression or death (whatever occurs first).
  patients with platinum-sensitive recurrent ovarian cancer with a positive AGO Score
Quality of Life measures with EORTC QLQ-C30 Global Health Status (GHS) | Baseline, 6, and 12 months after randomization
  GHS scale-core item 29, 30; ranges 0-100
Quality of Life measures with EORTC QLQ-C30 Symptom Scale Insomnia | Baseline, 6, and 12 months after randomization
  Item 11, ranges 0-100
Quality of Life measures with EORTC QLQ-C30 Symptom Scale Constipation | Baseline, 6, and 12 months after randomization
  Item 16, ranges 0-100
Quality of Life measures with FACT-G total score | Baseline, 6, and 12 months after randomization
  Composite of 27 items regarding physical, functional, social/family and emotional well-being. from 0-108
Quality of Life measures with FACT-O Ovarian Cancer subscale | Baseline, 6, and 12 months after randomization
  Composite of 11 items regarding specific to Ovarian Cancer patients, ranges 0-44
Quality of Life measures with FACT-O total score | Baseline, 6, and 12 months after randomization
  Sum of FACT-G and and Ovarian Cancer subscale, ranges 0-152

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Harter, MD, Principal Investigator — AGO Study Group
Locations (86):
- Austria (4):
  - Medizinische Universität Graz, Universitätsklinik für Frauenheilkunde Graz, Abteilung Gynäkologie u. Geburtshilfe, Graz
  - Universitätsklinikum Innsbruck, Univ. Klinik für Gynäkologie und Geburtshilfe, Innsbruck
  - Medizinische Universität Wien,Universitätsklinik für Frauenheilkunde, Vienna
  - Wilhelminenspital der Stadt Wien, Gynäkologisch und Geburtshilfliche Abteilung, Vienna
- UZ Leuven, Leuven, Belgium
- China (4):
  - Zhejiang Cancer Hospital, Gynecology Oncology, Hangzhou
  - Fudan University Cancer Hospital, Gynecologic Oncology, Shanghai
  - Fudan University Zhongshan Hospital, Obstetrics and Gynecology, Shanghai
  - Suzhou Municipal Hospital, Gynecologic and Obstetrics, Suzhou
- Denmark (5):
  - Aalborg Hospital, Aalborg
  - Aarhus University Hospital,Oncology, Aarhus
  - Ringshospitalet Copenhagen University Hospital; Oncology, Copenhagen
  - Herlev Hospital, Herlev
  - Odense University Hospital, Gynaecology and Obstetrics, Odense
- France (12):
  - Institut Bergonié, Gynecology, Bordeaux
  - Centre Francois Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Antoine Lacassagne, Nice
  - Hôpital Européen Georges Pompidou, Paris
  - Hôpital Tenon, Paris
  - Insitut Jean Godinot, Service Rubis - Oncologie Médicale, Reims
  - Centre Eugène Marquis, Rennes
  - Centre Hospitalier Universitaire Charles-Nicolle, Rouen
  - Centre Henri Becquerel, Rouen
  - Centre René Gauducheau, Saint-Herblain
  - Centre Claudius Regaud, Toulouse
- Germany (25):
  - Hochtaunus-Kliniken gGmbH, Frauenklinik, Bad Homburg
  - Charité - Universitätsmedizin Berlin, Campus Virchow-Klinikum, Klinik für Frauenheilkunde, Berlin
  - Universitätsklinikum Carl Gustav Carus, Klinik für Frauenheilkunde u. Geburtshilfe, Dresden
  - Evangelisches Krankenhaus, Frauenklinik, Düsseldorf
  - Kaiserswerther-Diakonie, Florence-Nightingale Krankenhaus, Gynäkologie, Düsseldorf
  - Kliniken Essen Mitte, Evang. Huyssens-Stiftung, Gynäkologische Onkologie, Essen
  - Klinikum der JWG Universität Frankfurt, Klinik für Gynäkologie und Geburtshilfe, Frankfurt am Main
  - Universitätsklinikum Freiburg, Frauenklinik, Freiburg im Breisgau
  - Klinikum Fürth, Frauenklinik Nathanstift, Fürth
  - Georg-August-Universität Göttingen, Universitäts-Frauenklinik, Göttingen
  - Gynecologic Clinic of the Ernst-Moritz-Arndt-University, Greifswald
  - Medizinische Hochschule, Klinik für Frauenheilkunde u. Geburtshilfe, Hanover
  - Klinikum Kempten, Klinik für Frauenheilkunde und Geburtshilfe, Kempten
  - Universitätsklinikum Schleswig-Holstein Campus Kiel, Klinik f. Gynäkologie u. Geburtshilfe, Kiel
  - Klinikum Konstanz, Frauenklinik, Konstanz
  - Universitätsklinikum Schleswig-Holstein, Campus Lübeck, Klinik für Frauenheilkunde und Geburtshilfe, Lübeck
  - Universitätsklinikum Mainz, Frauenklinik, Mainz
  - Klinikum Dritter Orden, Gynäkologie und Geburtshilfe, München
  - Klinikum der Universität München-Großhadern, Klinik und Poliklinik für Frauenheilkunde und Geburtshilfe, München
  - Oberschwaben Klinik, Krankenhaus St. Elisabeth, Frauenklinik, Ravensburg
  - Caritas-Krankenhaus St. Josef, Klinik für Frauenheilkunde und Geburtshilfe d. Universität Regensburg, Regensburg
  - Leopoldina-Krankenhaus der Stadt Schweinfurt GmbH, Frauenklinik, Schweinfurt
  - Universitätsklinikum, Universitätsfrauenklinik, Ulm
  - Ammerland-Klinik GmbH, Frauenklinik, Westerstede
  - HSK, Dr. Horst Schmidt Klinik GmbH, Klinik für Gynäkologie u. Gynäkologische Onkologie, Wiesbaden
- Italy (4):
  - Centro di Riferimento Oncologico,Struttura Operativa complessa Chirurgia Oncologica Ginecologica, Aviano
  - Fondazione IRCCS Istituto Nazionale Tumori di Milano, Milan
  - Istituto Europeo di Oncologia, Divisione di Ginecologia, Milan
  - Istituto Nazionale Tumori di Napoli, Gynecologic Oncology, Naples
- Norwegian Radium Hospital, Oslo University Hospital, Gynecologic Oncology, Oslo, Norway
- Seoul National University Hospital, Department of Obstetrics and Gynecology, Seoul, South Korea
- Spain (9):
  - ICO Badalona - H. U. Germans Trias i Pujol, Badalona
  - Hospital de la Santa Creu i Sant Pau, Oncology, Barcelona
  - Hospital Clinic Barcelona, Oncology, Barcelona
  - ICO-Hospital Universitari de Girona Dr. Josep Trueta, Servicio de Oncologia de Girona, Girona
  - Avinguda Granvia de l'Hospitalet de Llobregat, Hospital de Bellvitge, Gynaecology, L'Hospitalet de Llobregat
  - Hospital Son Llàtzer, Oncology, Palma de Mallorca
  - Hospital de Navarra, Oncology, Pamplona
  - Fundación Instituto Valenciano de Oncologia, Valencia
  - Hospital Universitari i Politècnic la Fe, Oncology, Valencia
- Sweden (2):
  - Linköping University Hospital, Department of Obstetrics and Gynecology, Linköping
  - Karolinska University Hospital, Oncology, Stockholm
- United Kingdom (18):
  - Birmingham City Hospital, Cancer Research Team, Birmingham
  - Cambridge University Hospitals NHS FT - Addenbrookes Hospital, Gynaecological Oncology, Cambridge
  - Queen Elizabeth Hospital Gateshead, Northern gynaecological oncology centre, Gateshead
  - Royal Surrey Country Hospital,St Lukes Cancer Centre, Guildford
  - Lincoln County Hospital, Oncology, Lincoln
  - St Bartholomew´s Hospital and Queen´s Hospital,Gynaecological Cancer Centre, London
  - University College London Hospital, Cancer clinical trails unit, London
  - Royal Marsden NHS Foundation Trust, Gynae research, Mulberry House, London
  - Imperial College Healthcare NHS Trust Hammersmith Hospital, Medical Oncology, London
  - Central Manchester Foundation NHS Trust, St Mary´s Hospital, Gynaecology, Manchester
  - Queen Elizabeth the Queen Mother Hospital,East Kent Gynaeoncology Centre, Margate
  - Northampton General Hospital, Gynaecological Oncology, Northampton
  - East and North Hertfordhire NHS Trust,Mount Vernon Hospital,Medical Oncology, Northwood
  - Norfolk & Norwich University Hospital,Obstetrics & Gynaecology, Norwich
  - Nottingham University Hospital, City Campus, Oncology, Nottingham
  - Royal Hallamshire Hospital & Weston Park Hospital, Cancer Clinical Trials Centre, Sheffield
  - Princess Anne Hospital, gynaecology, Southampton
  - New Cross Hospital,Oncology/Gynaecology, Wolverhampton

REFERENCES:
- [Result] Harter P, Sehouli J, Vergote I, Ferron G, Reuss A, Meier W, Greggi S, Mosgaard BJ, Selle F, Guyon F, Pomel C, Lecuru F, Zang R, Avall-Lundqvist E, Kim JW, Ponce J, Raspagliesi F, Kristensen G, Classe JM, Hillemanns P, Jensen P, Hasenburg A, Ghaem-Maghami S, Mirza MR, Lund B, Reinthaller A, Santaballa A, Olaitan A, Hilpert F, du Bois A; DESKTOP III Investigators. Randomized Trial of Cytoreductive Surgery for Relapsed Ovarian Cancer. N Engl J Med. 2021 Dec 2;385(23):2123-2131. doi: 10.1056/NEJMoa2103294. PMID 34874631
- [Derived] Bommert M, Harter P, Heitz F, du Bois A. When should Surgery be used for Recurrent Ovarian Carcinoma? Clin Oncol (R Coll Radiol). 2018 Aug;30(8):493-497. doi: 10.1016/j.clon.2018.04.006. Epub 2018 May 7. PMID 29743148